

# TRIAL STATISTICAL ANALYSIS PLAN

c29131491-01

**BI Trial No.:** 1346-0029

**Title:** A study to investigate the effects of donepezil on the

pharmacokinetics of BI 425809 and vice versa in healthy male and female subjects (Open-label, two-treatment, two-period, one fixed

sequence cross-over design)

Including Protocol Amendment 3 [c26441921-04]

Investigational Product:

BI 425809

Responsible trial statistician:

Phone: Fax:

Date of statistical

**20 SEP 2019 SIGNED** 

analysis plan:

Version: Final


Proprietary confidential information

 ${\small ©~2019~Boehringer~Ingelheim~International~GmbH~or~one~or~more~of~its~affiliated~companies.~All~rights~reserved.}$ 

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

Boehringer Ingelheim
TSAP for BI Trial No: 1346-0029
Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### TABLE OF CONTENTS 1.

| TITLE | PAGE | 1 |
|------------|------------------------------------------------|----|
| 1. | TABLE OF CONTENTS | 2 |
| LIST O | OF TABLES | 4 |
| 2. | LIST OF ABBREVIATIONS | 5 |
| 3. | INTRODUCTION | 7 |
| 4. | CHANGES IN THE PLANNED ANALYSIS OF THE STUDY | |
| 5. | ENDPOINTS. | |
| 5.<br>5.1 | PRIMARY ENDPOINTS | |
| 5.1<br>5.2 | SECONDARY ENDPOINTS | |
| 5.2.1 | Key secondary endpoints | |
| 5.2.2 | Secondary endpoints | |
| 5.3.2 | Safety parameters | 9 |
| 5.4 | OTHER VARIABLES | |
| 5.4.1 | Demographic and other baseline characteristics | |
| 5.4.2 | Treatment compliance and treatment exposure | 10 |
| 6. | GENERAL ANALYSIS DEFINITIONS | |
| 6.1 | TREATMENTS | |
| <b>6.2</b> | IMPORTANT PROTOCOL DEVIATIONS | |
| 6.3 | SUBJECT SETS ANALYSED | 15 |
| 6.5 | POOLING OF CENTRES | 16 |
| 6.6 | HANDLING OF MISSING DATA AND OUTLIERS | |
| <b>6.7</b> | BASELINE, TIME WINDOWS AND CALCULATED VISITS | 16 |
| 7. | PLANNED ANALYSIS | 17 |
| 7.1 | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | 17 |
| 7.2 | CONCOMITANT DISEASES AND MEDICATION | |
| 7.3 | TREATMENT COMPLIANCE | |
| 7.4 | PRIMARY ENDPOINTS | |
| 7.4.1 | Primary analysis of the primary endpoints | 18 |
| 7.5 | SECONDARY ENDPOINTS | 19 |
| 7.5.1 | Key secondary endpoints | 19 |
| 7.5.2 | Secondary endpoints | 19 |
| 7.6.2 | Safety parameters | |
| 7.7 | EXTENT OF EXPOSURE | |
| <b>7.8</b> | SAFETY ANALYSIS | 20 |

# **Boehringer Ingelheim**

TSAP for BI Trial No: 1346-0029 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| <b>7.8.1</b> | Adverse Events | 20 |
|--------------|-----------------|----|
| 7.8.2 | Laboratory data | 21 |
| 7.8.3 | Vital signs | |
| 7.8.4 | ECG. | |
| 7.8.5 | Others | 22 |
| 10. | HISTORY TABLE | 26 |

# **Boehringer Ingelheim**

TSAP for BI Trial No: 1346-0029 
Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# LIST OF TABLES

| Table | 6.1: | l Dosage and treatment schedule part 1 | .11 |
|---|---|---|---|
| Table | 6.1: 2 | 2 Dosage and treatment schedule part 2 | .11 |
| Table | 6.1: 3 | Analysis phases for statistical analysis of AEs, vital signs, safety laboratory | |
| | | data and visual tests, part 1 | .12 |
| Table | 6.1: 4 | Analysis phases for statistical analysis of AEs, vital signs, safety laboratory | |
| | | data and visual tests, part 2 | .13 |
| Table | 6.2: | 1 Handling of IPDs | .15 |
| Table | 6.3: | Subject sets analyzed | .15 |
| Table | 10: 1 | History table | .26 |

Boehringer Ingelheim
TSAP for BI Trial No: 1346-0029 
Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 2. LIST OF ABBREVIATIONS

| Term | Definition / description |
|---|---|
| ADME | Absorption, Distribution, Metabolism and Excretion |
| AE | Adverse Event |
| AESI | Adverse event of special interest |
| ALT | Alanine aminotransferase |
| ANOVA | Analysis of variance |
| AST | Aspartate aminotransferase |
| $\mathrm{AUC}_{0	ext{-tz}}$ | Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point |
| $AUC_{0-\infty}$ | Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity |
| BI | Boehringer Ingelheim |
| BP | Blood pressure |
| $C_{\text{max}}$ | Maximum measured concentration of the analyte in plasma |
| CTP | Clinical Trial Protocol |
| CTR | Clinical Trial Report |
| CV | Arithmetic coefficient of variation |
| C-SSRS | Columbia Suicidal Severity Rating scale |
| ECG | Electrocardiogram |
| gCV | geometric coefficient of variation |
| gMean | Geometric mean |
| ICH | International Conference On Harmonisation |
| IPD | Important protocol deviations |
| IQRMP | Integrated quality and risk management plan |
| MedDRA | Medical Dictionary For Regulatory Activities |
| PK | Pharmacokinetics |
| PKS | Pharmacokinetic parameter set |
| PR | Pulse rate |
| RAGe | Report appendix generator |
| SAE | Serious adverse event |
| SD | Standard Deviation |
| SOC | System Organ Class |

# **Boehringer Ingelheim**

TSAP for BI Trial No: 1346-0029 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Term | Definition / description |
|------|---------------------------------|
| TS | Treated set |
| TSAP | Trial Statistical Analysis Plan |
| ULN | Upper limit of normal range |

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 3. INTRODUCTION

As per ICH E9 (1) the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the revised CTP, and to include detailed procedures for executing the statistical analysis of the primary variables and other data.

This TSAP assumes familiarity with the CTP and its amendments. In particular, the TSAP is based on the planned analysis specification as written in CTP Section 7 "Statistical Methods and Determination of Sample Size". Therefore, TSAP readers may consult the CTP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size, randomisation.

Study data will be stored in a trial database within Medidata Rave system.

The statistical analyses will be performed within the validated working environment CARE, including SAS<sup>TM</sup> (current Version 9.4, by SAS Institute Inc., Cary, NC, USA), and a number of SAS<sup>TM</sup>-based tools (e.g., macros for the analyses of AE data or laboratory data; Report Appendix Generator system (RAGe) for compilation/formatting of the CTR appendices).

PK parameters will be calculated using Phoenix WinNonlin<sup>TM</sup> software (version Phoenix 6.3, Certara USA Inc., Princeton, NJ, USA).

TSAP for BI Trial No: 1346-0029 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### CHANGES IN THE PLANNED ANALYSIS OF THE STUDY 4.

All analyses described in this TSAP are in accordance with the statistical methods described in the revised CTP.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 5. ENDPOINTS

#### 5.1 PRIMARY ENDPOINTS

Primary endpoints are PK endpoints of BI 425809 (part 1) and donepezil (part 2), as defined in Section 2.1.2 of the CTP:

- $AUC_{0-\infty}$  (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity)
- $C_{max}$  (maximum measured concentration of the analyte in plasma)

# 5.2 SECONDARY ENDPOINTS

# 5.2.1 Key secondary endpoints

Not applicable.

# 5.2.2 Secondary endpoints

Secondary endpoints are PK endpoints of BI 425809 (part 1) and donepezil (part 2), as defined in Section 2.1.3 of the CTP:

•  $AUC_{0-tz}$  (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point)

# **5.3.2** Safety parameters

Safety and tolerability of BI 425809 will be assessed based on further safety parameters defined in Section 2.2.2.2 of the CTP:

- Adverse events (including clinically relevant findings from the physical and neurological examination)
- Safety laboratory tests, including faecal occult blood test
- *12-lead ECG*
- Visual tests
- *Vital signs (blood pressure, pulse rate)*
- Suicidality assessment (C-SSRS, only part 2)

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 5.4 OTHER VARIABLES

# 5.4.1 Demographic and other baseline characteristics

**CTP:** At the screening visit, the medical examination will include documentation of subject information, informed consent, demographics including height and body weight, smoking and alcohol history, relevant medical history and concomitant therapy, review of inclusion and exclusion criteria, visual tests, C-SSRS assessment (only for Part 2), review of vital signs (BP, PR), 12-lead ECG, laboratory tests, and a physical examination (including a neurological examination consisting of Romberg and Unterberger test, assessment of gait, further tests as needed).

Body mass index will be calculated as weight [kg] / height [m]<sup>2</sup>.

# 5.4.2 Treatment compliance and treatment exposure

Treatment compliance will not be analysed as a specific endpoint, cf. Section 4.3 of the CTP.

Treatment exposure is defined as the total dose and number of doses of BI 425809 and donepezil per subject.

# 6. GENERAL ANALYSIS DEFINITIONS

### 6.1 TREATMENTS

For basic study information on treatments to be administered, assignment of treatment groups, and selection of doses, cf. Section 4 of the CTP.

Each subject is planned to be treated in two subsequent treatment periods in a fixed sequence order. There will be no washout-period between the two treatment periods.

#### Part 1:

All subjects will receive a single dose of BI 425809 alone in Visit 2 and a single dose of BI 425809 after multiple dosing of donepezil in Visit 3.

Table 6.1: 1 Dosage and treatment schedule part 1

| Treatment | Substance | Formulation | Unit<br>strength | Dosage | Total dose |
|---|---|---|---|---|---|
| A (Reference 1) | BI 425809 | Tablet | 25 mg | 1 tablet (Day 1, Visit 2) | 25 mg |
| B (Test 1) | Donepezil | Tablet | 5 mg | 1 tablet (Day 1-7, Visit 3) q.d.<br>2 tablets (Day 8-28, Visit 3) q.d. | 245 mg |
| | BI 425809 | Tablet | 25 mg | 1 tablet (Day 22, Visit 3) | 25 mg |

# Part 2:

All subjects will receive a single dose of donepezil alone in Visit 2 and then a single dose of donepezil after multiple dosing of BI 425809 in Visit 3.

Table 6.1: 2 Dosage and treatment schedule part 2

| Treatment | Culatora | Formulation | Unit | Dagage | Total daga |
|---|---|---|---|---|---|
| Treatment | Substance | romulation | strength | Dosage | Total dose |
| C (Reference 2) | Donepezil | Tablet | 5 mg | 2 tablets (Day 1, Visit 2) | 10 mg |
| D (Test 2) | BI 425809<br>Donepezil | Tablet<br>Tablet | 25 mg<br>5 mg | 1 tablet (Day 1-24, Visit 3) q.d.<br>2 tablets (Day 10, Visit 3) | 600 mg<br>10 mg |

For statistical analyses of AEs, vital signs, safety laboratory data and visual tests the following separate analysis phases will be defined for each subject:

Table 6.1: 3 Analysis phases for statistical analysis of AEs, vital signs, safety laboratory data and visual tests, part 1

| Study analysis | | | |
|---|---|---|---|
| phase | Label | Start | End |
| Screening | Screening part 1 | Date of informed consent | Date/time of first administration of BI 425809 |
| On treatment<br>BI 425809 | BI part 1 | Date/time of first administration of BI 425809 | Date/time of first administration of donepezil |
| On treatment donepezil | Don part 1 | Combination of two phases: | Combination of two phases: |
| donepozn | | First phase: Date/time of first administration of BI 425809 + 11*24h (i.e. REP of BI425809 of 11 days) | First phase:<br>Date/time of second<br>administration of BI 425809 |
| | | Second phase: Date/time of second administration of BI 425809 + 11*24h (i.e. REP of BI425809 of 11 days) | Second phase: Date/time of last administration of donepezil + 15*24h (i.e. REP of donepezil of 15 days) or 00:00 a.m. on day after subject's trial termination date whatever occurs earlier |
| On treatment BI 425809+ | Don + BI part 1 | Combination of two phases: | Combination of two phases: |
| donepezil | | First phase:<br>Date/time of first administration<br>of donepezil | First phase:<br>Date/time of first administration<br>of BI 425809 + 11*24h (i.e. REP<br>of BI425809 of 11 days) |
| | | Second phase:<br>Date/time of second<br>administration of BI 425809 | Second phase: Date/time of second administration of BI 425809 + 11*24h (i.e. REP of BI425809 of 11 days) |
| Follow-up | F/U part 1 | Date/time of last administration of donepezil + 15*24h (i.e. REP of donepezil of 15 days) | 00:00 a.m. on day after subject's trial termination date |

The planned duration of the analysis phase of BI part 1 is 8 days, of Don part 1 it is 28 days and of Don + BI part 1 it is 14 days.

Table 6.1: 4 Analysis phases for statistical analysis of AEs, vital signs, safety laboratory data and visual tests, part 2

| Study analysis phase | Label | Start | End |
|---|---|---|---|
| Screening | Screening part 2 | Date of informed consent | Date/time of first administration of Donepezil |
| On treatment donepezil | Don part 2 | Date/time of first administration of donepezil | Date/time of first administration of donepezil + 15*24h (i.e. REP of donepezil of 15 days) |
| On treatment BI 425809 | BI part 2 | Combination of two phases: | Combination of two phases: |
| 423009 | | First phase:<br>Date/time of first administration<br>of BI 425809 | First phase: Date/time of second administration of donepezil |
| | | Second phase: Date/time of second administration of donepezil + 15*24h (i.e. REP of donepezil of 15 days) | Second phase: Date/time of last administration of BI 425809 + 11*24h (i.e. REP of BI 425809 of 11 days) or 00:00 a.m. on day after subject's trial termination date |
| On treatment<br>BI 425809+<br>donepezil | BI + Don part 2 | Date/time of second administration of donepezil | whatever occurs earlier Date/time of second administration of donepezil + 15*24h (i.e. REP of donepezil of 15 days) |
| Follow-up | F/U part 2 | Combination of two phases: | Combination of two phases: |
| | | First phase: Date/time of first administration of donepezil + 15*24h (i.e. REP of donepezil of 15 days) | First phase:<br>Date/time of first administration<br>of BI 425809 |
| | | Second phase:<br>Date/time of last administration<br>of BI 425809 + 11*24h (i.e.<br>REP of BI 425809 of 11 days) | Second phase: 00:00 a.m. on day after subject's trial termination date |

The planned duration of the analysis phase of Don part 2 is 15 days, of BI part 2 it is 19 days and of BI + Don part 2 it is 15 days.

AE displays in CTR Section 15.3, Appendix 16.1.13.1.8.2 and Appendix 16.1.13.1.8.3 will present results for the on-treatment phase only.

In AE tables in CTR Section 15.3 (but not in Appendix 16.1.13.1.8.2 and Appendix 16.1.13.1.8.3 AE tables), the following total will be provided in addition:

- "Total on-trt part x", defined as the total over all on-treatment phases, x will be replaced with 1 or 2 for the respective part
- "Total BI part x", defined as the total over all on-treatment phases involving BI, x will be replaced with 1 or 2 for the respective part

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

CTR Appendix 16.1.13.1.8.1 displays will present results for the screening, on-treatment and follow-up phases.

Additionally to the total defined above, the following total will be provided in AE tables in CTR Section 16.1.13.1.8.1:

• "Total part x", defined as the total over all study phases (screening + on-treatment + follow-up), x will be replaced with 1 or 2 for the respective part

More details on the technical implementation of these analyses are provided in the ADS Plan of this TSAP.

# 6.2 IMPORTANT PROTOCOL DEVIATIONS

Consistency check listings (for identification of deviations from time windows) and a list of protocol deviations (e.g. deviations in drug administration, in blood sampling times, etc.) will be provided to be discussed at the Report Planning Meeting (RPM). At this meeting, it will be decided whether a discrepant data value can be used in analyses or whether it must be corrected in the clinical database. Each protocol deviation must be assessed to determine whether it is an important PD (IPD). For definition of IPDs, and for the process of identification of these, refer to the BI reference document "Identify and Manage Important Protocol Deviations (IPD)" (2).

If any IPDs are identified, they are to be summarised into categories and will be captured in the decision log. Categories that are considered to be IPDs in this trial are defined in the integrated quality and risk management plan (IQRMP). If the data show other IPDs, the definition in the IQRMP will be supplemented accordingly by the time of the RPM.

IPDs will be summarized and listed. <u>Table 6.2: 1</u> below specifies which kind of IPDs could potentially lead to exclusion from which analysis set. The decision on exclusion of subjects from analysis sets will be made at the latest at the RPM, after discussion of exceptional cases and implications for analyses. If the data show other IPDs, this table will be supplemented accordingly by the time of the RPM.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 6.2: 1 Handling of IPDs

| IPD code | IPD Category & Brief Description | Excluded from which analysis set |
|---|---|---|
| A1 | Inclusion Criteria Not Met | PKS |
| A2 | Exclusion Criteria Violated | PKS |
| B1 | Informed consent not available/not done | TS, PKS |
| B2 | Informed consent too late | None |
| C1 | Non-compliance | PKS |
| C2 | Incorrect intake of trial medication | PKS |
| СЗ | Incorrect trial medication taken | PKS |
| D1 | Prohibited medication use | PKS |
| D2 | Improper washout of prohibited concomitant medication | PKS |
| E1 | Certain violations of procedures used to measure primary or secondary data | PKS |
| F1 | Certain violations of time schedule used to measure primary or secondary data | PKS |
| G1 | PDs affecting safety and rights of subjects | None |

# 6.3 SUBJECT SETS ANALYSED

Subject sets will be used as defined in the CTP, Section 7.3.

Table 6.3: 1 Subject sets analyzed

| | Subj | ect set |
|----------------------------------------|------|---------|
| Class of endpoint | TS | PKS |
| Primary PK endpoints | | X |
| Secondary PK endpoints | | X |
| Safety parameters & treatment exposure | X | |
| Demographic/baseline | X | |
| endpoints | Λ | |

#### 6.5 POOLING OF CENTRES

This section is not applicable, because the study was performed in only one centre.

# 6.6 HANDLING OF MISSING DATA AND OUTLIERS

Data of screened subjects who were withdrawn from the trial prior to first administration of any study drug will not be reported in the CTR.

Data of subjects who failed to complete all periods of the study (dropouts or withdrawals) will be reported in the CTR as far as their data are available. All withdrawals will be documented and the reason for withdrawal reported in the CTR.

**CTP**: *It is not planned to impute missing values for safety parameters.* 

One exception where imputation might be necessary for safety evaluation are AE dates. Missing or incomplete AE dates are imputed according to BI standards ( $\underline{3}$ ).

Missing data and outliers of PK data are handled according to BI standards (4) and (5).

**CTP**: *PK* parameters that cannot be reasonably calculated based on the available drug concentration-time data will not be imputed.

# 6.7 BASELINE, TIME WINDOWS AND CALCULATED VISITS

Baseline is defined as the last available value before first drug administration.

Time windows are defined in Section 6.1 of the CTP. Adherence to time windows will be checked at the RPM.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 7. PLANNED ANALYSIS

The format of the listings and tables will follow the BI guideline "Reporting of clinical trials and project summaries" (6).

The individual values of all subjects will be listed. Listings will be sorted by treatment group subject number and visit (if visit is applicable in the respective listing). AE listings will be sorted by assigned treatment (see <u>Section 7.8.1</u> below for details). The listings will be contained in Appendix 16.2 (SDL) of the CTR.

The following standard descriptive statistical parameters will be displayed in summary tables of continuous variables:

N number of non-missing observations

Mean arithmetic mean SD standard deviation

Min minimum Median median Max maximum

For plasma concentrations as well as for all PK parameters the following descriptive statistics will additionally be calculated:

CV arithmetic coefficient of variation

gMean geometric mean

gCV geometric coefficient of variation

For PK parameters the following descriptive statistics will additionally be calculated:

P10 10<sup>th</sup> percentile Q1 1<sup>st</sup> quartile Q3 3<sup>rd</sup> quartile P90 90<sup>th</sup> percentile

The data format for descriptive statistics of plasma concentrations will be identical with the data format of the respective concentrations. The descriptive statistics of PK parameters will be calculated using the individual values with the number of decimal places as provided by the evaluation program. Then the individual values as well as the descriptive statistics will be reported with three significant digits in the CTR.

Tabulations of frequencies for categorical data will include all possible categories and will display the number of observations in a category as well as the percentage (%) relative to the respective treatment group. Percentages will be rounded to one decimal place. The category missing will be displayed if and only if there actually are missing values. Percentages will be based on all subjects in the respective subject set whether they have non-missing values or not.

#### 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Only descriptive statistics are planned for this section of the CTR.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7.2 CONCOMITANT DISEASES AND MEDICATION

Concomitant diseases will be coded according to the most recent version of MedDRA. Concomitant medication will be coded according to the most recent version of the World Health Organisation – Drug Dictionary. Concomitant non-drug therapies will be coded according to the most recent version of MedDRA.

A medication will be considered concomitant, if it

- is ongoing at the time of first study drug administration, or
- starts within the analysis phase of the respective treatment (see <u>Section 6.1</u> for a definition of treatments and analysis phases).

The relevance of the concomitant therapies to the evaluation of PK will be decided no later than at the RPM.

Only descriptive statistics are planned for this section of the CTR.

# 7.3 TREATMENT COMPLIANCE

Treatment compliance will not be analyzed as a specific endpoint. Any deviations from complete intake will be addressed in the Report Planning Meeting (cf. Section 6.2) and described in the CTR.

#### 7.4 PRIMARY ENDPOINTS

# 7.4.1 Primary analysis of the primary endpoints

Primary analysis of the primary endpoints will be performed as defined in Sections 7.3.1 of the CTP.

The statistical model for the primary analysis defined in the CTP is an analysis of variance (ANOVA) model on the logarithmic scale including "treatment" as fixed effects and "subject" as random effect. Relative bioavailability of the study treatments will be estimated by the ratios of the geometric means

- treatment B (Test 1)/treatment A (Reference 1) (part 1)
- treatment D (Test 2)/treatment C (Reference 2) (part 2)

of the primary endpoints.

# Exclusion of PK parameters

The ADS ADPP contains column variables APEXC and APEXCO indicating inclusion/exclusion (APEXC) of a PK parameter and an analysis flag comment (APEXCO). All analyses based on the PKS are based on PK parameter values which are not flagged for exclusion, i.e. with APEXC equal to "Included".

# Exclusion of plasma concentrations

The ADS ADPC (PK concentrations per time-point or per time-interval) contains column variables ACEXC or ACEXCO indicating inclusion/exclusion (ACEXC) of a concentration and an analysis flag comment (ACEXCO). Exclusion of a concentration depends on the analysis flag comment ACEXCO. For example, if ACEXCO is set to "ALL CALC", the value will be excluded for all types of analyses based on concentrations. If ACEXCO is set to "DESC STATS" the value will be excluded from descriptive evaluations per planned time point/time interval. If ACEXCO contains the addition "TIME VIOLATION" or "TIME DEVIATION", the value can be used for further analyses based on actual times. If ACEXCO is set to "HALF LIFE", the value will be excluded from half-life calculation only; the value is included for all other analyses. Excluded concentration itself will be listed in the CTR associated with an appropriate flag.

Further details are given in "Noncompartmental Pharmacokinetic / Pharmacodynamic Analyses of Clinical Studies" (4) and "Description of Analytical Transfer Files and PK/PD Data Files" (5).

# 7.5 SECONDARY ENDPOINTS

# 7.5.1 Key secondary endpoints

This section is not applicable as no key secondary endpoint has been specified in the protocol.

# 7.5.2 Secondary endpoints

The secondary endpoints will be statistically analysed in the same way as for the primary endpoints. The endpoints will also be assessed descriptively. The analysis of standard PK parameters is performed according to BI standards (4).

See <u>Section 7.4</u> of this TSAP for details regarding exclusion of PK parameters and plasma concentrations.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 7.6.2 Safety parameters

Safety endpoints and tolerability will be analysed as described in <u>Section 7.8</u> of this TSAP.

#### 7.7 EXTENT OF EXPOSURE

Descriptive statistics are planned for this section of the report.

#### 7.8 SAFETY ANALYSIS

All safety analyses will be performed on the TS.

### 7.8.1 Adverse Events

AEs will be coded with the most recent version of MedDRA.

The analyses of AEs will be descriptive in nature. All analyses of AEs will be based on the number of subjects with AEs and not on the number of AEs.

For analysis, multiple AE occurrence data on the eCRF will be collapsed into one event provided that all of the following applies:

- All AE attributes are identical (lower level term, intensity, action taken, therapy required, seriousness, reason for seriousness, relationship, outcome, AESI)
- The occurrences were time-overlapping or time-adjacent (time-adjacency of two occurrences is given if the second occurrence started at most 1 hour after the first occurrence ended)

For further details on summarization of AE data, please refer to "Analysis and Presentation of Adverse Event Data from Clinical Trials" (7) and "Handling of missing and incomplete AE dates" (3).

The analysis of AEs will be based on the concept of treatment emergent AEs. That means that all AEs will be assigned to screening, on-treatment or follow-up phases as defined in <a href="Section 6.1">Section 6.1</a>. AEs will be analysed based on actual treatments, as defined in <a href="Table 6.1:3">Table 6.1:3</a> and <a href="Table 6.1:4">Table 6.1:4</a>.

An overall summary of AEs will be presented. This overall summary will comprise summary statistics for the class of other significant AEs according to ICH E3 (8) and for the class of AESIs.

**CTP:** *The following are considered as AESIs:* 

- *Hepatic injury* 
  - A hepatic injury is defined by the following alterations of hepatic laboratory parameters:
  - $\circ$  An elevation of AST (aspartate transaminase) and/or ALT (alanine transaminase)  $\geq 3$ -fold ULN combined with an elevation of total bilirubin  $\geq 2$ -fold ULN measured in the same blood sample, or
  - $\circ$  Aminotransferase (ALT, and/or AST) elevations  $\geq$ 10 fold ULN

The investigator had to classify on the eCRF whether an observed AE was an AESI or not.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

According to ICH E3 (8) AEs classified as "other significant" need to be reported and will include those non-serious and non-significant AEs

- (i) which are marked haematological or other lab abnormalities, or
- (ii) which were reported with "action taken = discontinuation" or "action taken = reduced", or
- (iii) which lead to significant concomitant therapy as identified by the Clinical Monitor/Investigator at a Medical Quality Review Meeting.

The frequency of subjects with AEs will be summarised by treatment, primary SOC and preferred term. AEs which were considered by the investigator to be drug related will be summarised separately. Separate tables will also be provided for subjects with SAEs, subjects with AESIs and subjects with other significant AEs (according to ICH E3 (8)). AEs will also be summarized by maximum intensity.

The SOCs and preferred terms within SOCs will be sorted by descending frequency over all treatment groups.

For disclosure of AE data on ClinicalTrials.gov, the frequency of subjects with non-serious AEs occurring with an incidence of greater than 5 % (in preferred terms) will be summarised by treatment, primary SOC and preferred term. The frequency of subjects with SAEs will also be summarised.

For disclosure of AE data in the EudraCT register, the frequency of AEs, the frequency of non-serious AEs with an incidence of greater than 5 % (in preferred terms) and the frequency of SAEs will be summarized.

For support of lay summaries, the frequency of subjects with drug-related SAEs will be summarized by treatment, primary SOC and preferred term.

# 7.8.2 Laboratory data

The analyses of laboratory data will be descriptive in nature and will be based on BI standards "Display and Analysis of Laboratory Data" (9).

Analyses will be based on normalised values, which means transforming to a standard unit and a standard reference range. The original values will be analysed if the transformation into standard unit is not possible for a parameter.

Descriptive statistics of absolute values and change from baseline from laboratory parameters over time (see <u>Section 6.7</u>) will be provided. Frequency tables of changes between baseline and last value on treatment with respect to the reference range will be presented.

Unscheduled measurements of laboratory data will be assumed to be repeat measurements of the most recent scheduled measurement (e.g. for follow-up or confirmation of a particular value). Therefore, unscheduled measurements will be assigned to the planned time point of the previous scheduled measurement. Descriptive statistics will be calculated by planned time point based on the worst value of the subject at that planned time point (or assigned to that planned time point).

Possibly clinically significant abnormal laboratory values are only those identified either in the Investigator's comments or at the RPM at the latest. It is the Investigator's responsibility to decide whether a lab value is clinically significant abnormal or not. Standard or project-

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

specific rules for flagging clinically significant values in an automated manner will not be applied in this study.

Clinically relevant findings in laboratory data will be reported as baseline conditions (prior to first administration of study treatment) or as AEs (after first administration of study treatment) if judged clinically relevant by the investigator, and will be analyzed as such.

Results from the fecal occult blood testing will be listed only.

### 7.8.3 Vital signs

The analyses of vital signs (blood pressure and pulse rate) will be descriptive in nature. Descriptive statistics of absolute values and change from baseline from vital signs over time (see Section 6.7) will be provided.

Unscheduled measurements of vital signs will be assigned to planned time points in the same way as described above for laboratory data. However, for vital signs, descriptive statistics will be calculated by planned time point based on the last value of the subject at that planned time point (or assigned to that planned time point).

Clinically relevant findings in vital signs data will be reported as baseline conditions (prior to first administration of study treatment) or as AEs (after first administration of study treatment) if judged clinically relevant by the investigator, and will be analyzed as such.

#### 7.8.4 ECG

Relevant ECG findings will be reported as relevant medical history/baseline condition (if a condition already exists before first administration of study treatment) or as AE (if condition emerges after first administration of study treatment) and will be summarized as such. No separate listing or analysis of ECG findings will be prepared.

## **7.8.5** Others

Physical and neurological examination findings will be reported as relevant medical history/baseline condition (if a condition already exists before first administration of study treatment) or as AE (if condition emerges after first administration of study treatment) and will be summarized as such. No separate listing or analysis of physical or neurological examination findings will be prepared.

# **Suicidality assessment**

Suicidality monitoring will be performed as described in Section 5.2.4 of the CTP, results will only be listed. No further analysis will be prepared. Findings will also be reported as AEs.

# Visual test

Visual test will be performed as described in Section 5.2.3 of the CTP.

Unscheduled measurements of visual tests will be assigned to planned time points in the same way as described above for laboratory data. However, for visual tests, descriptive statistics

will be calculated by planned time point based on the last value of the subject at that planned time point (or assigned to that planned time point).

# Colour discrimination test

Abnormal findings during the screening examination will lead to exclusion of the subject. Any deterioration during the study compared to baseline will be reported as an AE. Results from all measurements will also be listed and summarized in a frequency table for each eye.

# Visual acuity test

Any deterioration during the study compared to baseline will be reported as an AE. Results from all measurements will be listed and summarized including change from baseline separately for each eye.

# Amsler grid test

Abnormal findings during the screening examination will lead to exclusion of the subject. Any deterioration during the study compared to baseline will be reported as an AE. Results from all measurements will also be listed and summarized for each eye.

TSAP for BI Trial No: 1346-0029 
Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

TSAP for BI Trial No: 1346-0029 
Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# **Boehringer Ingelheim**

TSAP for BI Trial No: 1346-0029 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **10. HISTORY TABLE**

Table 10: 1 History table

| Version | Date<br>(DD-MMM-YY) | Author | Sections changed | Brief description of change |
|---|---|---|---|---|
| Final | 20-SEP-2019 | | None | This is the final TSAP |